CLINICAL TRIAL: NCT07149688
Title: Village-Based Management of Chronic Cardiovascular Disease in Qu Jiang Elderly Population Registry: The BOUQUET Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: The BOUQUET Cohort Study
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF); Hypertension; Coronary Heart Disease (CHD); Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Coronary Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Comprehensive management program (pharmacologic treatment, lifestyle modification, health education, structured follow-up) — Comprehensive management program (pharmacologic treatment, lifestyle modification, health education, structured follow-up)
  Enhanced monitoring with 7-day ECG

SUMMARY:
This is a prospective observational cohort study conducted in Qujiang District, Zhejiang Province, China, aiming to evaluate the effectiveness of a comprehensive management program for elderly patients with chronic cardiovascular diseases (CVDs). The program integrates pharmacological treatment, lifestyle modification, health education, and long-term follow-up, with enhanced monitoring using 7-day ECG recording. The study focuses on major chronic CVDs including hypertension, coronary artery disease, atrial fibrillation, and heart failure. Approximately 30,000 participants aged ≥60 years will be enrolled and followed for up to 10 years.

DETAILED DESCRIPTION:
With the acceleration of global population aging, older adults have become the primary population at high risk for chronic cardiovascular diseases (CVD). Cardiovascular disease is one of the leading causes of mortality and disability worldwide, and its prevalence and associated disability are markedly higher among the elderly compared to younger age groups. According to data from the World Health Organization (WHO), CVD accounts for approximately 31% of global deaths, with older adults carrying a substantial proportion of this burden.

Due to age-related physiological changes, the presence of multiple comorbidities, and lifestyle factors, elderly individuals often face more complex health challenges. In this population, chronic hypertension, coronary artery disease, heart failure, and diabetes are highly prevalent and frequently coexist. These conditions tend to be chronic, progressive, and involve multiple organ systems, further complicating disease management. Moreover, elderly patients often experience poor drug tolerance, multiple complications, and impaired quality of life, which necessitate not only more refined clinical interventions but also individualized management strategies tailored to patient-specific needs.

Traditional single-disease treatment strategies are often insufficient to address the multifaceted needs of elderly patients with chronic cardiovascular diseases. Existing evidence suggests that comprehensive management models-integrating multidisciplinary collaboration, personalized treatment, long-term follow-up, and health education-can significantly improve cardiovascular outcomes, reducing hospitalization rates, mortality, and other adverse events. However, systematic research on comprehensive management in elderly populations remains limited. Most current studies focus on specific diseases or therapeutic approaches, lacking multidimensional assessment and intervention strategies.

Therefore, the present study aims to establish a comprehensive management cohort for chronic cardiovascular diseases in elderly populations, in order to explore how integrated management strategies influence cardiovascular health in real-world settings. This study will evaluate the effectiveness of such approaches in reducing cardiovascular events and mortality, thereby providing scientific evidence and guidance for future clinical practice. The Qujiang Project Team of the National Clinical Research Center for Cardiovascular Diseases will undertake this study.

ELIGIBILITY:
Inclusion Criteria

Age ≥60 years

Resident of Qujiang District

Diagnosed with chronic CVD (hypertension, coronary artery disease, heart failure, atrial fibrillation, or others)

Able and willing to provide informed consent

Exclusion Criteria

Severe cognitive impairment or inability to provide consent

Life expectancy <1 year due to non-cardiovascular disease

Participation refusal

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling elderly residents of Qujiang District with chronic cardiovascular diseases.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2035-03-01 (Estimated); Study Completion 2035-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events | 10 years
  Incidence of cardiovascular events (myocardial infarction, stroke, hospitalization for heart failure, cardiovascular death) - assessed annually during follow-up
All-cause and cardiovascular mortality | 10 years
  All-cause and cardiovascular mortality - assessed at 10 years

SECONDARY OUTCOMES:
Hospitalization rates | 10 years
  Hospitalization rates (number and duration of hospitalizations for CVD-related causes)
Atrial fibrillation burden | 10 years
  Atrial fibrillation burden - time proportion of AF episodes, number of episodes, longest episode duration (measured during 7-day ECG monitoring in the blanking period and annually thereafter)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No